CLINICAL TRIAL: NCT05302570
Title: PROTONS-RPS: a Phase II Non-Randomized Open-label Single-arm Trial Of Neoadjuvant Short-course Hypofractionated Proton Beam Therapy for Non-metastatic RetroPeritoneal Sarcoma
Brief Title: Neoadjuvant Short-course Hypofractionated PBT for Non-metastatic RPS
Acronym: PROTONS-RPS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: withdrawn by PI
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Robert L. Sloan Fund for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00315399
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Retroperitoneal Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated Proton Beam Therapy (Experimental): 5 fractions of 5 Gy of PBT to clinical tumor volume +/- an additional simultaneous 1 Gy per fraction to any pre-determined at-risk margin (for a total of 6 Gy per fraction x 5 fractions for at-risk margins as a simultaneous integrated boost (SIB)).
  Interventions: Radiation: Hypofractionated Proton Beam Therapy

INTERVENTIONS:
Radiation: Hypofractionated Proton Beam Therapy — 5 fractions of 5 Gy of PBT to clinical tumor volume +/- an additional simultaneous 1 Gy per fraction to any pre-determined at-risk margin (for a total of 6 Gy per fraction x 5 fractions for at-risk margins as a simultaneous integrated boost (SIB)).

SUMMARY:
The investigators' study titled "PROTONS-RPS: a Phase II non-Randomized Open-label single-arm Trial Of Neoadjuvant Short-course hypofractionated proton beam therapy for non-metastatic RetroPeritoneal Sarcoma" is a phase II trial evaluating the safety and efficacy of hypofractionated proton beam therapy (H-PBT) in the neoadjuvant (NA) setting for patients with non-metastatic retroperitoneal sarcoma (RPS) planned for surgical resection. This trial will include adult patients with resectable RPS.

DETAILED DESCRIPTION:
The investigators' primary outcome is overall complication rate after treatment with NA H-PBT and surgical resection based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.2 Secondary objectives include evaluating the acute toxicity of H-PBT prior to surgical resection, rate of progression between diagnosis and definitive resection, early post-operative complication rate after resection of RPS in patients who received NA H-PBT, and local recurrence-free survival at 1 and 2 years. A priori subset analyses will be conducted for patients with well-differentiated and dedifferentiated liposarcoma.

The investigators plan to accrue a minimum of 44 patients to evaluate the investigators' primary outcome. Treatment will be 5 doses of H-PBT including a simultaneous integrated boost to at-risk margins followed by surgical resection after 4-6 weeks. Patients will be followed in the post-operative setting according to standard of care surveillance for RPS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age)
* Patients with primary non-recurrent retroperitoneal sarcoma
* Calculated creatinine clearance ≥50 mL/min and functional contralateral kidney based on nuclear medicine renal scan
* Normal bone marrow function (WBC ≥ 4 x109 /L)
* Eastern Cooperative Oncology Group status ≤ 2
* Cardiac function ≤ New York Heart Association class II
* Proton beam therapy approved by insurance (including Medicare/Medicaid)

Exclusion Criteria:

* Evidence of metastatic disease on staging CT of chest/abdomen/pelvis
* History of abdominal or pelvic radiation therapy
* Inability to tolerate supine position for duration of PBT simulation or treatment
* Tumor originating from gastrointestinal or gynecologic organs
* Specific sarcoma histologies including osteosarcoma, desmoid tumors, chondrosarcoma arising from vertebrae or pelvic bones, embryonal rhabdomyosarcoma
* Tumor extending into femoral or obturator canal
* History of systemic lupus erythematosus or ulcerative colitis
* Genetic syndrome with radiation-associated tumorigenicity (i.e.: Li-Fraumeni)
* Presence of clinically significant ascites
* Co-existing malignancy or treated malignancy in the last 2 years expected to limit life expectancy; does not include completely resected cutaneous basal cell carcinoma, squamous cell carcinoma, in situ breast or cervical malignancies, or other pathologies at the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall serious adverse event rate for patients with primary resectable RPS receiving NA short-course h-PBT followed by surgical resection | 24 months
  Incidence of acute Grade 3+ adverse events after PBT and surgical resection during median follow-up based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Safety of NA short-course hypofractionated PBT for primary resectable RPS as assessed by incidence of acute Grade 3+ adverse events | Up to 6 weeks
  Safety determined by incidence of acute Grade 3+ adverse events per the NCI CTCAE v5.0 in patients on treatment with H-PBT prior to surgical resection.
Tolerability of NA short-course hypofractionated PBT for primary resectable RPS as assessed by cessation of NA H-PBT due to toxicity or required dose reduction for serious adverse events | Up to 6 weeks
  Lack of tolerability determined by cessation of NA H-PBT due to toxicity or required dose reduction for serious adverse events (NCI CTCAE v5.0).
Rate of local or distant tumor progression from diagnosis to time of surgery after treatment with PBT | Up to 6 weeks (pre-operatively)
  Local or distant tumor progression based on RECIST 1.1 criteria on pre-operative contrast-enhanced CT scan of the chest, abdomen, and pelvic compared to staging CT.
Rate of acute post-operative surgical complications in patients receiving NA short-course hypofractionated PBT | 30 days after surgery
  Incidence of 30-day (acute) post-operative complications based on Clavien-Dindo classification.
Local recurrence-free survival (LRFS) | Every 6 months, Up to 2 years
  Time from study enrollment to the earliest of local recurrence, death, or loss to follow-up after NA short-course h-PBT and resection. Recurrence will be determined on CT of the thorax, abdomen, and pelvis at 6-month intervals for 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Amol Narang, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No